CLINICAL TRIAL: NCT07216807
Title: Randomized Trial of Text vs. Video Patient Educational Materials in Cirrhosis
Brief Title: EDUCATE-C: Education on Cirrhosis -- Assessing Text vs Video
Acronym: EDUCATE-C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Patricia Bloom, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00204958
Record Dates: First submitted 2025-09-29; First posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- General cirrhosis text (Other): These patients received TEXT education, and the subject was general cirrhosis knowledge.
  Interventions: Other: Text education
- General cirrhosis video (Other): These patients received VIDEO education, and the subject was general cirrhosis knowledge.
  Interventions: Other: Video Education
- Decompensation text (Other): These patients received TEXT education, and the subject was decompensated cirrhosis knowledge.
  Interventions: Other: Text education
- Decompensation video (Other): These patients received VIDEO education, and the subject was general cirrhosis knowledge.
  Interventions: Other: Video Education

INTERVENTIONS:
Other: Video Education — Video education was provided from the cirrhosis.ca website.
  Arms: Decompensation video; General cirrhosis video
Other: Text education — Text education was provided from the University of Michigan patient education materials
  Arms: Decompensation text; General cirrhosis text

SUMMARY:
A randomized controlled trial of written text vs video education to patients with cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosis

Exclusion Criteria:

* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-20 (Actual)

PRIMARY OUTCOMES:
Delta knowledge scores between text and video education groups | Baseline and immediately post-intervention (Day 1)
  The delta score (post test minus pre test) was compared between text education and video education groups.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT07216807/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/07/NCT07216807/ICF_001.pdf